CLINICAL TRIAL: NCT06605027
Title: Therapeutic Ketogenic Diet to Treat Anorexia Nervosa-Specific Cognitions and Behaviors - Currently Ill Individuals in PHP Level of Care and Comparison With Standard of Care
Brief Title: Therapeutic Ketogenic Diet in Partial Hospital Program (PHP) Anorexia Nervosa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 810945
Record Dates: First submitted 2024-09-06; First posted 2024-09-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Subjects will be given the option to participate in the study intervention or continue to receive standard of care treatment in a structured high level of care eating disorders program.
Masking Description: Subjects will be able to choose which arm they participate in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic Ketogenic Diet (TKD) Study Arm (Experimental): Participants in the TKD Study Arm will complete 14 weeks of therapeutic ketogenic diet (TKD), weekly weight and ketone measurements, weekly behavioral assessments, and meetings with the study doctor and dietician every week, and peer counseling sessions.
  Interventions: Other: Therapeutic Ketogenic Diet
- Treatment as Usual (TAU) Study Arm (No Intervention): Participants who consent to be in the Treatment as Usual Study Arm will complete weekly weight and ketone measurements and questionnaires for 14 weeks.

INTERVENTIONS:
Other: Therapeutic Ketogenic Diet — 2 week induction to establish ketosis followed by 12 weeks therapeutic ketogenic diet
  Arms: Therapeutic Ketogenic Diet (TKD) Study Arm

SUMMARY:
This will be a 14-week longitudinal study with an open design. A total of 120 individuals will be recruited for an end goal of 60 individuals with anorexia nervosa (AN) who are currently in high level of care treatment at the UCSD Eating Disorder Center partial hospital program (PHP) or intensive outpatient (IOP). Forty individuals will be recruited to the TKD and 20 will be treated with treatment as usual with respect to food intake. The age range will be between 16 and 45 years. All study participants will be carefully assessed and will complete rater and self-assessments at the being at the end of the study period. While in the treatment program, the TKD group will receive catered ketogenic meals via a meal service. After discharging from program, participants will have the option to continue with the meal service or cook for themselves. After establishing ketosis, study participants will continue TKD for 12 weeks. All study participants will be followed over three, six, and twelve months after enrolling in the study, whether initiating TKD or being in the treatment as usual arm. This follow-up procedure will help determine whether symptom improvement is stable or worsens in individuals who choose to continue or discontinue the TKD intervention and in relation to the control group. After ketosis induction over two weeks, study participants will be assessed weekly for ketosis and mood, anxiety, and eating disorder symptoms over twelve weeks.

DETAILED DESCRIPTION:
For this 14-week study, 60 individuals with anorexia nervosa (AN) who are currently in high level of care treatment at the UC San Diego Health Eating Disorders Center for Treatment and Research (UC San Diego Health EDC) partial hospitalization program (PHP) or IOP will be recruited. These individuals will be underweight or recently weight-restored and continue to have high impairment from the illness as indicated by an Eating Disorder Examination Questionnaire (EDE-Q) global score greater than 2.09.

Of those 60 participants, 40 of them will participate in the Therapeutic Ketogenic Diet (TKD) Study Arm and 20 subjects will be enrolled in the Treatment as Usual Study Arm. The study will be conducted in a university medical environment, showing feasibility and safety in a typical medical setting.

After completing the screening steps all participants will complete a blood draw and genetics testing.

AN subjects will be given the option to participate in the TKD Study Arm or the Treatment as Usual Study Arm. Recruitment in each arm will continue until the end recruitment enrollment goal for each arm has been reached. Subjects will not be randomized to the study arm and will be given a choice of what arm they want to participate in. Subjects who consent to be in the TKD Study Arm will complete 14 weeks of therapeutic ketogenic diet (TKD), weekly weight and ketone measurements, weekly behavioral assessments, and meetings with the study doctor and dietician every week, and peer counseling sessions. While in the treatment program, the TKD group will receive catered ketogenic meals via a meal service. After discharging from program, participants will have the option to continue with the meal service or cook for themselves.

AN subjects who consent to be in the Treatment as Usual Study Arm will complete weekly weight and ketone measurements and questionnaires for 14 weeks.

After discharge from the PHP program, subjects will continue to be monitored virtually for the study procedures.

In the last week of the therapeutic ketogenic diet (week 14), all AN subjects will complete another blood draw and the exit visit with the study doctor and dietician.

AN subjects will complete follow-up visits 3 months, 6 months, and 1 year after the 14-week completion date.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form/parental permission form
2. Provision of signed and dated assent form if the subject is a minor
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Persons, aged 16 to 45 years
5. Current anorexia nervosa diagnosis according to DSM-5 criteria
6. An elevated EDE-Q global score of 2.09 or greater
7. The following types of psychiatric medications are allowed: antidepressant, anxiolytic, atypical antipsychotic, mood stabilizers
8. English is primary spoken language

Exclusion Criteria:

1. Pregnancy or lactation
2. Electrolyte, blood count, kidney function or liver function abnormalities
3. Psychosis
4. Neurocognitive disorders including dementias or traumatic brain injury that is symptomatic
5. Current alcohol use disorder (AUD) or substance use disorder (SUD) according to DSM-5 criteria
6. Uncontrolled hypertension
7. Hepatic impairment (Class-Pugh b or c)
8. Diabetes mellitus
9. Family history of porphyria
10. History of recent heart attack, vascular disease, or any other current acute medical conditions as determined by the principal investigator
11. Inability or unwillingness to adhere to the TKD diet for the duration of the study
12. Blind or illiterate individuals

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability in individuals with anorexia nervosa who are in a high level of eating disorder treatment using weekly body weight measurements. | Weekly for the duration of the study intervention (14 weeks)
  Weekly weights will be obtained to assess whether subjects remain within the clinical goal weight range.
To assess the safety and tolerability in individuals with anorexia nervosa who are in high level of eating disorder treatment using the Committee of Clinical Investigations UKU-Side Effect Scale (UKU Side Effect Rating Scale) | At weeks 4, 8, 12
  The UKU Side Effect Rating Scale assesses psychic, neurologic, autonomic, and other side effects on a scale of 0 to 3 where 0 = not or doubtfully present, 1 = present to a mild degree, 2 = present to a moderate degree, 3 = present to a severe degree. The global score ranges from 0 to 48 where a higher score indicates more side effects of the study intervention.
Measurement of drive for weight loss, fear of weight gain and body image distortion using the Eating Disorder Examination Questionnaire (EDEQ) Global Score | At baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 3 month follow-up, 6 month follow-up, 1 year follow-up
  The Eating Disorders Examination Questionnaire a self report assessment that measures core eating disorder symptoms. Subjects will complete this measure at the beginning and end of the study and weekly throughout the 14-week intervention and the investigator will measure the change in scores. The EDE Global scale has a range of 0 to 6 where higher scores mean worse outcome.
Measurement of drive for weight loss, fear of weight gain and body image distortion using the Eating Disorder Examination Questionnaire (EDEQ) Eating Restraint Score | At baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 3 month follow-up, 6 month follow-up, 1 year follow-up
  The Eating Disorders Examination Questionnaire a self report assessment that measures core eating disorder symptoms. Subjects will complete this measure at the beginning and end of the study and weekly throughout the 14-week intervention and the investigator will measure the change in scores. The EDE Restraint scale has a range of 0 to 6 where higher scores mean worse outcome.
Measurement of drive for weight loss, fear of weight gain and body image distortion using the Eating Disorder Examination Questionnaire (EDEQ) Weight Concern Score | At baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 3 month follow-up, 6 month follow-up, 1 year follow-up
  The Eating Disorders Examination Questionnaire a self report assessment that measures core eating disorder symptoms. Subjects will complete this measure at the beginning and end of the study and weekly throughout the 14-week intervention and the investigator will measure the change in scores. The EDE Weight concern scale has a range of 0 to 6 where higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calabrese L, Scolnick B, Zupec-Kania B, Beckwith C, Costello K, Frank GKW. Ketogenic diet and ketamine infusion treatment to target chronic persistent eating disorder psychopathology in anorexia nervosa: a pilot study. Eat Weight Disord. 2022 Dec;27(8):3751-3757. doi: 10.1007/s40519-022-01455-x. Epub 2022 Aug 23. PMID 35997954
- [Background] Dignon A, Beardsmore A, Spain S, Kuan A. 'Why I won't eat': patient testimony from 15 anorexics concerning the causes of their disorder. J Health Psychol. 2006 Nov;11(6):942-56. doi: 10.1177/1359105306069097. PMID 17035265
- [Background] Frank GKW, Shott ME, DeGuzman MC. The Neurobiology of Eating Disorders. Child Adolesc Psychiatr Clin N Am. 2019 Oct;28(4):629-640. doi: 10.1016/j.chc.2019.05.007. Epub 2019 Jul 4. PMID 31443880
- [Background] Scolnick B, Zupec-Kania B, Calabrese L, Aoki C, Hildebrandt T. Remission from Chronic Anorexia Nervosa With Ketogenic Diet and Ketamine: Case Report. Front Psychiatry. 2020 Jul 30;11:763. doi: 10.3389/fpsyt.2020.00763. eCollection 2020. PMID 32848935